# Lactate Kinetics Analysis Related to Low-Intensity Resistance

# **Exercise: Randomized Control Trial**

# 3 Abstract

- 4 Background: Virtual reality exercise (VRE) has been proven to overcome fatigue in hospital
- 5 setting. However, no study analyzes how lactate, as fatigue biomarker, is affected by VRE.
- 6 This study aims to analyze lactate kinetics as an exercise response after conventional
- 7 multimodal exercise and virtual reality exercise (VRE) in hospitalized geriatric.
- 8 Methods: Sixty subjects were randomized into control and VRE group. VRE is given as
- 9 adjuvant therapy to conventional multimodal exercise. Peripheral blood lactate was taken
- immediately before and after low-intensity resistance exercise at baseline and one week after.
- 11 The comparison of lactate changes between groups was analyzed using the Mann-Whitney
- 12 test.
- 13 Results: There is no difference in post-exercise lactate at day 1 and 7 between the two groups.
- Lactate concentrations reduce after low-intensity resistance exercise in subjects with high
- resting lactate -0.4(-0.45 0.5) but remain escalated in the normal group 0.1(-1 3.9) at day
- 16 1, p < 0.001.
- 17 Conclusion: There is no significant effect of VRE as an adjuvant therapy on post-exercise
- lactate. The next study needs to consider elevated baseline lactate to reduce bias. Also, the
- intensity of resistance exercise needs to be improved to high intensity through individual
- 20 exercise test.
- 21 Keywords: Exercise, Geriatric, Lactate, Virtual Reality

### Introduction

1

Advanced technology development of Virtual Reality (VR) has brought it from community 2 utilization into the hospital setting. VR has been used in a broad spectrum of diseases and 3 health conditions as part of prevention, promotive, curative, and rehabilitation strategies.<sup>2,3,4</sup> 4 Adaptation of VR in specific populations, such as children and the elderly, makes it more 5 popular as an advanced technology alternative in clinical settings.<sup>3,5</sup> VR allows patients and 6 7 medical team explore beyond hospital walls, thus enriching the medical management. Fatigue is a clinical symptom that commonly found in the elderly. It brings geriatric 8 syndromes and lead to disability. Fatigue has been proven to be effectively managed by VR. 9 VR effects on fatigue were dramatic and satisfaction. Fatigue was significantly decreased in 10 VR group while almost no changes were observed in control group. <sup>7,8</sup> Few of the studies even 11 proved that fatigue improves within 2 days after VR.<sup>9</sup> 12 VR activity had to be adjusted to the targeted disease or health condition. Actually, the 13 pathophysiology of fatigue involves two main organs: brain and muscle. 10 Some biomarkers 14 are also involved in fatigue, the most important are serotonin and lactate. 10,11 Previous study 15 might be addressed VR intervention in one of organs and biomarkers involved in fatigue. VR 16 that targeting brain and serotonin was designed as distraction intervention during unpleasant 17 protocol such as chemotherapy or hemodialysis.<sup>7,8</sup> The distraction hopefully could divert 18 subject's focus and enhance copying mechanism. VR that targeting muscle and lactate was 19 designed as virtual reality exercise (VRE).9 As principle of exercise, VRE must induced 20 physical activity. VRE must improve muscle performance, qualitative and quantitative. 21 Unfortunately, all of previous VR studies measure fatigue using scale or questionnaires, 22 could not directly prove the involvement of those organs and biomarkers. This study aims to 23 analyze lactate kinetics as an exercise response after conventional multimodal exercise and 24 VRE in hospitalized geriatric. 25

### 1 METHODS

# 2 Subject

- 3 Sixty geriatric patients were recruited during their hospitalization at RSUPN Dr. Cipto
- 4 Mangunkusumo (RSCM). As per description, subjects categorized as geriatric patients are
- 5 not only because their age is more than 59 years old, but also because they have multiple
- 6 comorbidities and geriatric syndromes. Subject was included if they able to communicate and
- 7 their manual muscle test results are minimal 3. They were excluded if they had VR-sickness,
- 8 severe psychosocial problem, and severe caregiver burden. They considered drop out if they
- 9 were discharged, worsen clinical condition and death before finishing the research protocol.

### 10 Study design

16

23

- Subjects were randomized into control and intervention group. Both groups get conventional
- multimodal exercise, the intervention group gets additional VRE as adjuvant therapy. Due to
- the nature of the exercise, the research was single blind. This study was registered in Health
- Research Ethical Committee, Faculty of Medicine, Universitas Indonesia, RSCM. Number of
- ethical approval letter is ND-47/UN2.F1/ETIK/PPM.00.02/2025.

#### **Conventional Multimodal Exercise**

- Exercise protocol that is given during hospitalization had been standardized and approved as
- 18 RSCM clinical practice guideline. Exercise prescription was given after the subjects going
- 19 through functional assessment conducted by physiatrists. The prescription described the
- 20 frequency, intensity, interval, and type of exercise that is adjusted to subject's clinical
- 21 condition. Each subject could have more than one type of exercise, but the most common
- combination consists of breathing, resistance, and aerobic exercises.

### Virtual Reality Exercise

- VRAGMENT software was administered as VRE to the intervention group. VRAGMENT is
- an abbreviation of Virtual Reality for Cognitive and Dementia. It was innovated in 2022 by

- 1 Universitas Indonesia through the collaboration of Indonesian Medical Education and
- 2 Research Institute (IMERI), Physical Medicine & Rehabilitation (PM&R) Department and
- 3 Industrial Engineering Department. VRAGMENT runs on the Oculus Meta Quest 2<sup>®</sup>. In
- 4 VRAGMENT, subjects should make phone call, groceries and making payment. Those
- 5 activities in virtual environment initiated real movement of neck, trunk, arms, and legs.

# 6 Lactate Kinetic Measurement

- 7 Capillary blood lactate sample was examined using StatStrip® from Nova Biomedical.
- 8 Measurement range of StatStrip<sup>®</sup> is 0,3 20,0 mmol/L. Lactate examination conducts at
- 9 baseline and one week after the exercise program. Blood samples were collected immediately
- pre and post-standardized low-intensity resistance training.

### 11 Statistical Analysis

- 12 The data collected were analyzed using SPSS statistics (version 24.0). Demography and
- clinical data were presented in mean (standard deviation), or median (minimum maximum),
- or proportion in percentage. The difference of lactate kinetics between group was analyzed
- using Mann-Whitney test.

# 1 RESULTS

- 2 Subject's characteristics between groups were homogenous. Mean age of subjects was 68
- 3 years, and most of them were male. Main diagnosis proportion was almost same between
- 4 both groups, as described in table 1. The five most common diagnoses in both groups were
- 5 Neoplasm, Hepatitis, Pneumonia, Cholangitis, and Gastroenteritis.

# 6 Table 1. Subject's Characteristic

| | Control $(n = 29)$ | VRE (n=32) | p |
|-------------------------|--------------------|--------------|-------|
| Age, $\overline{x}(SD)$ | 68,31 (5,90) | 68,06 (5,53) | 0,866 |
| Gender | | | 0,723 |
| Male, n (%) | 15 (51,7) | 18 (56,3) | |
| Main Diagnosis, n (%) | | • | 0,581 |
| Hepatitis | 7 (24,1) | 2 (22,2) | |
| Pneumonia | 4 (13,8) | 5 (15,6) | |
| Cellulites | 2 (6,9) | 2 (6,3) | |
| Neoplasm | 8 (27,6) | 11 (34,4) | |
| SLE | Ó | 1 (3,1) | |
| Cholangitis | 4 (13,8) | 5 (15,6) | |
| Gastroenteritis | 3 (10,3) | 2 (6,3) | |
| Fracture | Ó | 2 (6,3) | |
| Nephrolithiasis | 0 | 1 (3,1) | |
| Heart Failure | 1 (3,4) | 1 (3,1) | |

<sup>7</sup> VRE = Virtual Reality Exergame

- 8 There is no difference in post-exercise lactate in day 1 and 7 between groups, as describe in
- 9 Table 2.

# 10 Table 2. Post-Exercise Lactate Between Study Groups

| <b>Post-Exercise Lactate</b> | Control | VRE | р |
|------------------------------|----------------|----------------|-------|
| Day 1 | 1,6 (0,6 -3,3) | 1,5(0,6-4,2) | 0,882 |
| Day 7 | 1,4(0,4-3,6) | 1,6 (0,6 -5,5) | 0,123 |
| $\Delta$ Day 1 to 7 | 0.0(-1.5-1.9) | 0.0(-1.5-2.7) | 0,923 |

- 11  $\Delta$  Day 1 to 7 = Post-Exercise lactate Day 1 Post-Exercise lactate Day
- The pattern pre and post exercise lactate at day 1 and 7 was described in figure 1S. Higher
- post-exercise lactate than pre-exercise was found only in VRE group at Day 7.



2 Figure 1. Pre and Post-exercise lactate between control and VRE group in day 1 and day 7.

- 3 An analytical study of the effect of pre-exercise elevated lactate is presented in Table 2.
- 4 There was a significant difference of post-exercise lactate between subjects with normal and
- 5 elevated pre-exercise lactate at day 1.

6 Table 3. Post-exercise lactate based on baseline resting lactate concentration at Day 1

| Post Evanoisa I actata | Resting Lactate Concentration at Day 1 | | p |
|---|---|---|---|
| Post- Exercise Lactate | Normal | Elevated | |
| Day 1 | 1,3 (0,6 – 4,2) | 2,3 (0,6 – 3,6) | 0,001* |
| Day 7 | 1,3(0,4-3,9) | 1,7(0,6-5,5) | 0,124 |
| Δ Day 1 to 7 | 0.0(-1.5-1.4) | 0.1(-1.5-2.7) | 0,205 |

- Δ Day 1 to 7 = Post-Exercise lactate Day 1 Post-Exercise lactate Day 7. \* shows statistically
  significant, p<0,05.</li>
- 9 As described in Figure 2, if we look deeper in those subjects with elevated resting lactate at
- Day 1, both the control and the VRE groups showed a consistent decrease in post-exercise

- 1 lactate levels in Day 7 compare to Day 1. The decreased in VRE group seemed to be lower
- than the control group.



Figure 2. Post-exercise lactate between control and VRE group in day 1 and day 7.

### DISCUSSION

1

This study did not demonstrate the significance of the VRE effects on lactate kinetics (Table 2 3 2.). However, this study could describe the lactate kinetics of conventional training and VRE, particularly in the subgroup with elevated resting lactate levels on day 1 (Table 3. and Figure 4 2.). The decrease in post-exercise lactate on day 7 compared to day 1 indicates that the 5 subjects were becoming more trained, and muscle performance was improving. 6 7 Previous study had proven that routine exercise with fixed load, after a certain period, does not statistically influence resting blood lactate concentrations; however, it might decrease the 8 post-exercise lactate concentrations.<sup>12</sup> In that study, the Standardized Mean Difference 9 (SMD) was 0,73 mmol/L decreased from baseline. That is obviously different from this 10 study, which remained unchanged. The difference is most likely caused by the relatively 11 short observation interval in this study, which is 1 week, while in the previous study it was 12 12 weeks. 13 14 Another factor that may cause lactate not to change within 1 week, is an acute lactate response that does not align with the physiological pattern. Physiologically, the average 15 concentration of blood lactate after resistance training increases compared to baseline, with a 16 sequential average of 0.94(0.38) to 1.58(0.54) mmol/L.<sup>13</sup> In this study, the physiological 17 responses were only observed in the intervention group during the evaluation period, as 18 shown in Figure 1. 19 This may be caused by the symptom-limited resistance exercise methods that was applied to 20 the subjects. In this method, exercise would be terminated when the subject was fatigue and 21 cannot continue the exercise. In normal or trained subjects, this condition would occur when 22 the lactate threshold (LT) is exceeded. 14 leading to fatigue. In this study, the subjects had 23 various conditions that could affect fatigue. The main diagnoses of subjects were dominated 24

with infection and inflammatory diseases. Those might lead to premature exercise due to 1 fatigue arising from various uncontrolled factors in this research. 10 2 3 Another possible cause was the disruption of glycogenolysis metabolic function. Glycogenolysis is an anaerobic metabolism process in which glycogen is converted into ATP. 4 occurring in the liver, muscles, and adipose tissue. Previous studies have shown that subjects 5 with glycogenolysis disorders significantly experience an increase in lactate uptake after 6 exercise for several minutes, leading to a decrease in blood lactate levels. 15 In contrast, the 7 control group experiences an increase in lactate production, resulting in higher blood lactate 8 9 levels. Glycogenolysis impairment can occur due to genetic diseases or increased insulin activity. Insulin stimulates the body to meet its needs through aerobic metabolism, while 10 concurrently increasing Protein Phosphatase I (PPI), which ultimately reduces 11 glycogenolysis. This aerobic metabolism will also increase lactate uptake as one of the fuels 12 for aerobic metabolism. 16 Considering that hepatitis is one of the 5 most common diseases 13 14 (Table 1.), glycogenolysis disorders in the majority of subjects in this study might had occurred. 15 This study presents protocol and analysis for single-blinded randomized control trial 16 analyzing the effect of VRE in managing fatigue. Previous studies have proven that VRE was 17 effective in managing fatigue, 1,17 but this study advances for some reasons. The VRE used 18 VRAGMENT, which was designed in Bahasa and Indonesian culture. The groceries in the 19 virtual market were local brands. Payment in the virtual market was also using Indonesian 20 virtual money. Fatigue was measured with lactate, which responded immediately after 21 resistance exercise. This could control the effect of others such as infection and 22 inflammation, that might appear during hospitalization and affect lactate concentration (Table 23 1). Also, the control group of this study had standard inpatient exercises, not untreated group 24 as previous study. Standard inpatient exercises had proven to manage fatigue. 18 The last 25

- 1 reason was geriatric as the target population. Geriatric already well known prone to fatigue
- 2 since they had multiple comorbidities.
- 3 Lactate kinetics is a concept to simulate models of lactate production and removal from
- 4 blood. Some factors may induce lactate kinetics, one of them is exercise. After exercise,
- 5 blood lactate concentration remains improved as glycogenolysis happens, at the beginning of
- 6 exercise and after aerobic threshold exceeded. Lactate removal as exercise respond could take
- 7 place as lactate reuptake by muscle to be utilized as aerobic metabolism fuel. 19
- 8 The descriptive data shows that one week of conservative multimodal exercises could reduce
- 9 post-exercise lactate, Table 2. It may conclude that subjects got used to training and
- underwent less fatigue than at baseline, though the reduction was not statistically or clinically
- 11 significant.<sup>12</sup>
- On the other hand, the VRE group shows physiological lactate kinetics on day 7, Figure 1.
- 13 This indicated that the resistance exercise intensity that was performed fulfilled the overload
- principle. The overload principle refers to the concept of gradually increasing the intensity,
- duration, or frequency of exercise. This is important to stimulate fitness improvement.<sup>20</sup>
- Unfortunately, the important finding above did not meet the criteria for statistical and clinical
- significance. However, the descriptive data suggest that VRE has potential in enhancing
- 18 conservative exercise to meet the overload exercise principle.
- 19 Since lactate concentration in this study is still affected by elevated resting lactate (Table 3
- and Figure 3), the next study needs to consider elevated baseline lactate to reduce bias. Also,
- 21 the intensity of resistance exercise needs to be improved to high intensity through an
- 22 individual exercise test.

# **1 Conflicts of Interest**

- 2 The authors confirm no conflict of interest in this study
- **3 Funding Sources**
- 4 None
- 5 Acknowledgment
- 6 None

### REFERENCES

- 2 1. Ioannou A, Papastavrou E, Avraamides MN, Charalambous A. Virtual reality and
- 3 symptoms management of anxiety, depression, fatigue, and pain: a systematic review.
- 4 Vol. 6, SAGE Open Nursing. Nicosia: SAGE Publications Inc.; 2020. p. 1–13.
- 5 2. BR K, MH C, LS K, JY P. Effect of Virtual Reality on Cognition in Stroke Patients.
- 6 Ann Rehabil Med. 2011;35(4):450–9.
- 7 3. A. Suharti, M. Harini, L. Arif, N. Valentina BA. Safety Aspect of VR-based IADL
- 8 Rehabilitation Program for Elderly Patient: A Pilot Study. Jakarta; 2023.
- 9 4. Vlake JH, Bommel J Van, Wils EJ, Korevaar TIM, Hellemons ME, Schut AFC, et al.
- Effect of intensive care unit-specific virtual reality (ICU-VR) to improve
- psychological well-being and quality of life in COVID-19 ICU survivors: a study
- protocol for a multicentre, randomized controlled trial. Trials. 2021;22:328.
- 13 5. Wang EY, Kennedy KM, Zhang L, Qian D, Forbes T, Zuniga-Hernandez M, et al.
- Predicting pediatric healthcare provider use of virtual reality using a technology
- acceptance model. JAMIA Open. 2023;6(3):12–5.
- 16 6. Patino-Hernandez D, David-Pardo DG, Borda MG, Pérez-Zepeda MU, Cano-Gutiérrez
- 17 C. Association of fatigue with sarcopenia and its elements: a secondary analysis of
- SABE-Bogotá. Gerontol Geriatr Med. 2017;3:1–7.
- 7. Schneider SM, Hood LE. Virtual reality: A distraction intervention for chemotherapy.
- 20 Oncol Nurs Forum. 2007;34(1):39–46.
- 8. Schneider SM, Prince-Paul M, Allen MJ, Silverman P, Talaba D. Virtual reality as a
- distraction intervention for women receiving chemotherapy. Oncol Nurs Forum.
- 23 2004;31(1):81–8.
- 24 9. Cho H, Sohng KY. The effect of a virtual reality exercise program on physical fitness,
- body composition, and fatigue in hemodialysis patients. J Phys Ther Sci.

- 1 2014;26:1661–5.
- 2 10. Borren NZ, van der Woude CJ, Ananthakrishnan AN. Fatigue in IBD: epidemiology,
- pathophysiology and management. Vol. 16, Nature Reviews Gastroenterology and
- 4 Hepatology. Rotterdam: Nature Publishing Group; 2019. p. 247–59.
- 5 11. Beneke R, Leithsuser RM. Lactate metabolism. In: Encyclopedia of Exercise Medicine
- in Health and Disease. Berlin: Springer Berlin Heidelberg; 2012. p. 501–36.
- 7 12. Zhao T, Le S, Freitag N, Schumann M, Wang X, Cheng S. Effect of chronic exercise
- 8 training on blood lactate metabolism among patients with type 2 diabetes mellitus: a
- 9 systematic review and meta-analysis. Front Physiol. 2021;12:1–13.
- 10 13. Nitzsche N, Schulze R, Weigand F, Hummer N, Schulz H. Comparison of an acute
- resistance training on the lactateconcentration with and without blood flow restriction
- at different loads. Dtsch Z Sportmed. 2018;69:337–43.
- 13 14. Goodwin ML, Harris JE, Hernández A, Gladden LB. Blood lactate measurements and
- analysis during exercise: a guide for clinicians. J Diabetes Sci Technol. 2007;1:558–
- 15 69.
- 16 15. Hsieh WM, Chen CC, Wang SC, Tan SY, Hwang YS, Chen SC, et al. Virtual reality
- system based on kinect for the elderly in fall prevention. Technol Heal Care.
- 18 2014;22:27–36.
- 19 16. Vavřička J, Brož P, Follprecht D, Novák J, Kroužecký A. Modern perspective of
- lactate metabolism. Physiol Res. 2024;9973:499–514.
- 21 17. Cortés-Pérez I, Sánchez-Alcalá M, Nieto-Escámez FA, Castellote-Caballero Y,
- Obrero-Gaitán E, Osuna-Pérez MC. Virtual reality-based therapy improves fatigue,
- 23 impact, and quality of life in patients with multiple sclerosis. A systematic review with
- 24 a meta-analysis. Sensors. 2021;21(21):1–21.
- 18. Jung MW, Wallek S, Senn-Malashonak A, Schubert P, Siegler K, Rosenhagen A, et al.

- Effects of a structured exercise therapy on cancer-related fatigue during and after
- 2 paediatric stem cell transplantation: a randomized controlled trial. Physiother Q.
- 3 2021;29(3):76–85.
- 4 19. Stallknecht B, Vissing J, Galbo H. Lactate production and clearance in exercise.
- 5 Effects of training. A mini-review. Scand J Med Sci Sport. 1998;8(3):127–31.
- 6 20. American College of Sport Medicine. ACSM's guidelines for exercise testing and
- prescription. 11th ed. Liguori G, Feito Y, Fountaine C, Roy BA, editors. Philadelphia:
- 8 Walters Kluwer; 2022.

9